CLINICAL TRIAL: NCT04296721
Title: Cost-effectiveness Study of an Integrated Tertiary Hospital-primary Care Lifestyle Change Program for the Treatment of Obstructive Sleep Apnea Syndrome and Obesity
Brief Title: Cost-effectiveness Study of a Lifestyle Change Program for the Treatment of OSA and Obesity: Hospital-Primary Care.
Acronym: SPP-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Neus Salord Oleo, Medical Doctor, PH D, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR 229/17
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Obstructive Sleep Apnea of Adult; Obesity; Lifestyle; Weight Loss
Keywords: Obstructive sleep apnea; Obesity; Weight loss program; Exercise; CPAP treatment
MeSH Terms: conditions — Obesity; Weight Loss; Sleep Apnea, Obstructive; Motor Activity

STUDY DESIGN:
Intervention Model Description: Controled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive weight-loss program (Experimental): The life style change program will consist of two stages. The first will consist of a 3-month period of intensive diet and progressive exercise with biweekly consultations with a nutritionist (in groups or individually). The second stage will last for 9 months, until completion, with a diet that is progressively higher in calories, with more intense exercise, under the supervision of a community nurse and an individual nutritional consultation at 9 months.
  Interventions: Behavioral: Intensive weigh-loss program
- Standard dietary recommendations (Active Comparator): Patients will be followed according to the usual recommendations: A written diet (designed by a hospital nutritionist) and an exercise plan, depending on the patient's age and activity level, without any other type of evaluation or visit Visits in the Sleep Disorders Unit will be scheduled at 3 and 12 months
  Interventions: Behavioral: Standard Dietary recommendations

INTERVENTIONS:
Behavioral: Intensive weigh-loss program — Intervention group: Intensive weight-loss program: 0-3 months very low calorie diet, 15 days substituting three meals for low calorie shakes, from 15 to 120 days substituting 1 meal and from 120 days to 12 months on a low calorie diet while starting a progressive exercise programme. Recommendations for good sleep habits will be given. The program will be carried out through group and individual sessions with the hospital dietician. After 3 months: group sessions with a nurse in the basic area. Group sessions led by hospital dietician. From 3 to 12 months: group sessions led by primary care nurse.
  Arms: Intensive weight-loss program
Behavioral: Standard Dietary recommendations — Patients will be managed according to the usual recommendations: The common written diet (designed by a hospital nutritionist) and an exercise advice will be given according to patient age and level of activity, without any other assessment or additional visits.
  Arms: Standard dietary recommendations

SUMMARY:
Obesity is the main risk factor for Obstructive Sleep Apnea (OSA). Nasal CPAP is the standard treatment for OSA, but since weight-loss programs are not usually offered to OSA patients, the root causes of their illness and its comorbidities are not treated. There is some evidence regarding improvements in OSA after weight reduction but whether weight reduction programs are cost-efficient has not as yet been addressed. OBJECTIVE: To determine whether an intensive weight-loss program, carried out in a project combining hospital and primary care levels, is cost-effective in the medium and long term for the treatment of obese patients with severe OSA undergoing CPAP treatment. More concretely, our objective is to demonstrate whether this program achieves sufficient improvement in OSA to allow a reduction <30/h in the apnea-hypopnea index in at least 25%, improving their metabolic profile and central obesity. METHOD: A prospective, randomized, controlled study. Control group: standard dietary recommendations.

Intervention group: 0-3 months very low calorie diet, 15 days substituting three meals for low calorie shakes, from 15 to 120 days substituting 1 meal and from 120 days to 12 months on a low calorie diet while starting a progressive exercise program. Recommendations for good sleep habits will be given. The program will be carried out through group and individual sessions with the hospital dietician. After 3 months: group sessions with a nurse in the basic area. Group sessions led by hospital dietician. From 3 to 12 months: group sessions led by primary care nurse. MEASUREMENTS: At the beginning, at 3 and at 12 months: two-night home respiratory polygraph, actigraphy, anthropometric and blood analysis data including metabolic syndrome and inflammatory markers, and health related quality of life questionnaires. Direct and indirect costs of treatments, outpatient's consultations, incomes, emergency visits and patients' travel costs to medical centers.

DETAILED DESCRIPTION:
HYPOTHESIS The implementation of an intensive weight loss program, initiated under the supervision of an expert nutritionist and continued under the supervision of a trained primary care nurse can help obese patients with severe obstructive sleep apnea (OSA) undergoing continuous positive airway pressure (CPAP) treatment to achieve significant weight loss and will result in a reduction in OSA severity in a significant percentage of patients leading to the possibility of their ceasing CPAP treatment.

The program will also improve the control of comorbidities, hypertension, diabetes and dyslipidemia and inflammation.

OBJECTIVES

Primary objective Assess whether a lifestyle change program, carried out in a combined and coordinated way with the hospital and primary care environments, can be cost-effective in the medium and long term for the treatment of OSA in obese patients with severe OSA who are already receiving CPAP treatment. In particular, to demonstrate that the program is able to achieve sufficient improvement in OSA to provide at least 25% of patients with a reduction of apnea hypopnea index (AIH <30/h).

Secondary objectives Assess whether a lifestyle change program in obese patients with OSA who are already receiving CPAP treatment can achieve lower blood pressure levels, improve blood lipids and glycemic control and reduce C reactive protein and central obesity.

Assess the OSA improvement predictor factors of an OSA improvement associated with weight loss.

STUDY SETTING:

The study will be performed at a tertiary hospital Sleep Unit and the Department of Endocrinology and Nutrition, and 5 primary care centers in the area of influence of the hospital. A community nurse and a referring physician will be selected at each center.

The study has been approved by the hospital's Ethics Committee. All participants will give their informed written consent.

All the study variables will be collected at baseline and the lifestyle change program will begin for patients in the treatment arm. Patients in the control group will continue with their regular visits. At three months and at one year after the beginning of treatment, sleep studies will be performed again and all of the other variables will be recorded for all of the patients. In order to prevent control group drop outs, at the end of the study, patients from the control group will invited to join the lifestyle change program.

Sample size estimation is based on comparing the percentage of patients that meet the primary outcome definition (patients who achieve an apnea hypopneas index (AHI) under 30 apneas-hypopneas per hour after 12 months of intervention) in two randomized groups. In the literature, no effect beyond 5% in AHI reduction has been observed with a regular dietary recommendation. So, in the control group, the expected percentage of patients that will meet the primary outcome is 2%. Kuna et al (Sleep 2013 36(5):64) observed a reduction in AHI to under 30 apneas-hypopneas per hour in 50% of patients undergoing an intensive diet intervention. In the investigators' context, with a severe population with a higher AHI at baseline, the investigators expect to reduce the apnea-hypopnea index (AHI) to under 30 apneas-hypopneas per hour in 25 % of patients undergoing the intervention.

Therefore, 90 patients (45 in each group) are required in order to have an 80% chance of detecting an increase in the primary outcome measure from 2% in the control group to 25% in the experimental group, with a significance of 5%. This estimation takes into account a dropout rate of 10%. The investigators will use an uncorrected chi-squared statistic to evaluate the null hypothesis that the primary outcome measures for experimental and control subjects are equal.

Lifestyle Change Program:

The life style change program will consist of two stages. The first will consist of a 3-month period of intensive diet and progressive exercise with biweekly consultations with a nutritionist (in groups or individually). The second stage will last for 9 months, until completion, with a diet that is progressively higher in calories, with more intense exercise, under the supervision of a community nurse. Five community nurses from the area of influence of our center will participate in a 6-hour course on nutrition and lifestyle interventions in which they will become familiarized with the educational materials used in primary care group visits. In the second stage, the group visits performed in primary care will reinforce the main hygienic-dietetic concepts introduced previously in the nutritionist sessions. After each group visit, a telephone meeting between the nutritionist and the community clinical nurse will be held to resolve doubts.

Diet: First Phase: 3 months.

* First 15 days: Very low calorie diet. A diet that is very low in calories will be started (600-800 Kcal, based on gender and level of physical activity) with low calorie shakes that will substitute the three main meals (breakfast, lunch and dinner) and the necessary food to make up the total calorie intake.
* Up to week 12: 1200 Kcal diet with a low calorie shake replacing dinner. Exercising begins. Every nutrition session will last from 60 to 90 minutes and will be conducted by a nutritionist.

The nutritionist will follow up on compliance with the program and monitor for potential adverse events at each visit. Also at each visit, the nutritionist will provide advice on diet and lifestyle, with a special emphasis on diet and exercise. Visits with the nutritionist will be biweekly group or individual. Group consultation will include 4 to 10 patients. (see Chart 1 attached).

At three months into the intervention, patients will be given dietary guidelines of 1200-1500 kcal. These will be adapted individually by the dietician according to the nutritional requirements estimated by applying the Mifflin-St Jeor/Harris Benedict, formula without the hypercaloric shake. Calories intake will be based on the Mediterranean diet with the following percentages of macronutrients: 15-20 % Proteins,44-55 % carbohydrates and a maximum of 35% lipids (<7% saturated fatty acids <7%, 15-20% monounsaturated fatty acids, <7% polyunsaturated faty acids according Spanish obesity society (SEEDO).

Second phase: 3 months to 1 year. Follow up at the Primary Health Centre (CAP) by a nursing team.Visits will take place every 1,5 months maintaining a group format in each center with an individual consultation with the nutritionist at 9 months.

The nurse responsible for the group will lead the group sessions in which the objectives of the treatment will be reinforced and will record patients' anthropometric data at each session.

Exercise Each training session will consist of stretching, 5-10' of warm-up (50-60% of the maximum HR), 40-50' of aerobic exercise performed at 70-80% of the maximum heart rate and 5-10 'of cooling down (50-60% of the maximum HR). The practice of at least 150 minutes / week of moderate activity according to World Health Organization (WHO) recommendations (World Recommendations on Physical Activity for Health WHO-Geneva 2009) will be advised. If during the exercise program there are musculoskeletal complaints that are considered relevant (an Visual Analog Scale for pain (VAS) score ≥4 on three consecutive occasions) they will be visited by the rehabilitation service. In order to promote the practice of physical exercise and the acquisition of this habit, Discounts will be offered for local municipal gyms that will offer adequate physical exercise programs for obese people, monitored by physiotherapists or technicians.

Control group: Patients will be managed according to the usual recommendations: The common written diet (designed by a hospital nutritionist) and an exercise advice will be given according to patient age and level of activity, without any other assessment or additional visits. Visits to the Sleep Disorders Unit will be scheduled to coincide with the assessments at 3 and 12 months, the same as for the intervention group.

Criteria for withdrawal from the study:

* Onset of osteoarticular pain that prevents a patient from continuing to exercise
* A patient's continued refusal to follow the recommended guidelines.

ETHICAL ISSUES: The study will be conducted in accordance with the principles of the Declaration of Helsinki, as well as of the Data Protection Act (Law 15/1999). All patients will be asked to provide informed consent, in accordance with the rules of the Ethics Committee at our institution. Since all of the patients will be receiving CPAP treatment, there should be no ethical concerns about evaluating the effectiveness of an alternative treatment that in principle is less effective than CPAP, in patients with severe OSA.

STATISTICAL ANALYSIS:

In order to evaluate the effectiveness of a change in lifestyle (diet and exercise) in obese patients with OSA, we will first perform a descriptive analysis of the demographic variables and baseline characteristics according to the number of cases and percentages for the qualitative variables and we will use measures of central tendency (mean, median) and dispersion (standard deviation and interquartile range) for the quantitative variables. In order to address the primary and secondary objectives of this study, we will run an inferential analysis comparing data at baseline, at 3 months and at one year in the two treatment groups. Tests for independent samples will be used in every case comparing the control and experimental groups). Either the chi-square test or Fisher's exact test will be used, as appropriate, to compare categorical variables and Student's T-test will be used to compare continuous variables; if the variable under study does not meet the conditions for the applicability of parametric tests, a non-parametric alternative, the Mann Whitney U test, will be used. An estimate of treatment effect in relation to the primary and secondary endpoints will be obtained from the confidence interval (95% CI) of the difference between means and percentages, as appropriate. The efficacy assessment will be based on an analysis of the per protocol populations (PP) and intention-to-treat (ITT), with the ITT population being the main analysis. For the population analysis using ITT, the missing data will be filled in and a sensitivity analysis will be conducted if more than one method of imputation is used. The PP population will be determined in accordance with compliance with visits, as well as with diet and exercise. A safety assessment will be made by identifying the adverse effects that are considered to be most significant due to their frequency or severity. In all cases, the significance level used will be 5% <0.05) with a bilateral approach. The statistical software used for the analysis will be IBM SPSS Statistics 21.

We will carry out two cost-effectiveness analyses, since we will use two effectiveness variables, The Short Form-36 Health Survey (SF-36) and the % decrease in AHI below 30, in the population studied in patients with severe OSA with a one-year follow-up. At first the database will be cleaned up and the cost allocation will be carried out by applying the flowchart. Then the analysis will determine the cost-effectiveness ratios (ICERs) acceptability curves, confidence ellipses and sensitivity analysis. A study of the costs will also be carried out taking into account the different hidden items.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with severe OSA (apnea apnea hypopnea index (AHI)> 30 / h),
* undergoing CPAP treatment for at least 6 months,
* with a body mass index (BMI)> = 30 kg / m2 y = <40 kg / m2,
* living in the area of the 5 participating primary care centers

Exclusion Criteria:

* diseases that can limit the practice of exercise or adherence to diet,
* severe cognitive or psychiatric disorders that prevent understanding of the program,
* serious illnesses, severe cardiovascular disease with clinical instability during the month prior to inclusion,
* prior bariatric surgery,
* refusal of the patient to participate in the study and craniofacial malformations that prevent OSA improvement.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Number of patients with Apnea Hypopnea Index under 30 per hour after receiving the program. Home Respiratory Polygraphy. | Baseline, at 3 months and 12 months
  Asses whether a lifestyle change program can be effective in medium and long term for treatment of OSA in obese OSA patients who are already receiving CPAP treatment.
Cost-effectiveness ot an intensive weight loss programme | Baseline, at 3 months and 12 months
  Asses whether a lifestyle change program can be cost-effective in medium and long term for treatment of OSA in obese OSA patients who are already receiving CPAP treatment.
Improvement of apnea-hypopnea index/hour: Home Respiratory polygraphy (Type 3) | Baseline, at 3 months and 12 months
  apnea-hypopnea index/hour: Home respiratory polygraphy (Type 3)
Direct and indirect costs | Baseline and 12 months
  All direct and indirect costs will be collected. Costs of CPAP and its fungibles, medical visits in primary care medicine and specialized medicine , hospital admissions and emergency consultations. Costs derived from sick leave. Costs derived from traffic and labor accidents. Costs of visits and tests carried out in the intervention. Cost derived of side effects from intervention. Patients Travel costs at the hospital and the primary medicine center. Costs derived from the use of sports equipment. Costs derived from side effects of the intervention. Mediation costs collecting changes during the protocol.

SECONDARY OUTCOMES:
Waist circumference | Baseline, at 3 months and 12 months
  Above the upper iliac crest: centimetre
Neck Circumference | Baseline, at 3 months and 12 months
  Neck Circumference: centimetre
Body fat Composition by bioimpedance analysis | Baseline, at 3 months and 12 months
  Body fat Composition by bioimpedance analysis (BIA 101, Akern Bioresearch, Florence, italy)
Measurement of health-related quality of life | Baseline, at 3 months and 12 months
  Questionnaire regarding quality of life: SF-36 Spanish language version SF-36 V1 Med Clin (Barc). 1995 May 27;104(20):771-6.
Cardiovascular risk factors and comorbidity | Baseline, at 3 months and 12 months
  Clinical questionnaire
Testing for Ketones | from baseline to 3 month.
  During very low diet to asses adherence to diet, testing for ketones using test strips will be performed.
Physical activity diary | Baseline, at 3 months and 12 months
  Record for physical activity (Weight loss program group)
Actigraphy | Baseline, at 3 months and 12 months
  Actiwattch Respironics monitoring system is going to be used to assess the subject's sleep/wake pattern and activity in response to therapy. Actigraphy Actiwath Respironics.. According to regulations of Spanish Sleep Society 2017 (ses.org.es).
Blood pressure | Baseline, at 3 months and 12 months
  Blood pressure measurement (BP) according to current spanish consensus guidelines (Gijón-Conde T, Hipertens Riesgo Vasc. 2018).
Fasting glucose | Baseline, at 3 months and 12 months
  Fasting glucose (millimol/liter)
weight | Baseline, at 3 months and 12 months
  weight Kg
Height | Baseline
  Height meters
Body Mass Index | Baseline, at 3 months and 12 months
  Dividing weight in kilograms by height in meters squared
Triglycerides (millimol/litter) | Baseline, at 3 months and 12 months
  fasting Triglycerides (millimol/litter)
Total Cholesterol | Baseline, at 3 months and 12 months
  Total fasting Cholesterol (millimole/liter)
Low Density lipoprotein (LDL) cholesterol (millimole/litter) | Baseline, at 3 months and 12 months
  Fasting Low Density lipoprotein (LDL) cholesterol (millimole/litter)
High Density lipoprotein (HLDL) cholesterol (millimole/litter) | Baseline, at 3 months and 12 months
  Fasting High Density lipoprotein (HLDL) cholesterol (millimole/litter)
Very Low lipoprotein (VLDL) cholesterol (millimole/litter) | Baseline, at 3 months and 12 months
  Fasting Very Low lipoprotein (VLDL) cholesterol (millimole/litter)
Glycosylated Hemoglobin | Baseline, at 3 months and 12 months
  Glycosylated Hemoglobin (5)
C-reactive protein (milligram/liter) | Baseline, at 3 months and 12 months
  serum C-reactive protein (milligram/liter)
Aspartate aminotransferase (microgram/liter) | Baseline, at 3 months and 12 months
  Aspartate aminotransferase (microgram/liter)
Alanine aminotransferase (microgram/liter) | Baseline, at 3 months and 12 months
  Alanine aminotransferase (microgram/liter)

OTHER OUTCOMES:
Self-perceived sleepiness | Baseline, at 3 months and 12 months
  Epworth Sleepiness score (MW Johns, Sleep 1991, 14; 540).
CPAP compliance | Baseline, at 3 months and 12 months
  hours of average night use from the hour meters. If there are patients that due to the
  weight loss, refer to intolerance to the pressure used, and need changes in pressure, changes will be collected or eventual suspension of the CPAP before the year of follow-up.
Visual Analog Scale for Pain (VAS) | Baseline, at 3 months and 12 months
  VAS Scale for Pain
Dietary questionaries | Baseline, at 3 months and 12 months
  In the intervention group adherence to diet wil be monitored by diet questionaries : 15-day dietary log and 24h Reminder log
Insulin (mUI / L) | Baseline, at 3 months and 12 months
  serum Insulin (mUI / L)
Homeostatic Model Assessment of Insulin Resistance. (HOMA-IR) | Baseline, at 3 months and 12 months
  Insulin resistance will be measured by HOMA-IR method [glucose (mmol / L) x insulin (mUI / L)] /22.5. d)

CONTACTS AND LOCATIONS:
Overall Officials: Neus Salord, MD, phD, Principal Investigator — Hospital Universitari de Bellvige
Locations (1):
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No